CLINICAL TRIAL: NCT00333489
Title: A National, Multicentric and Comparative Study to Evaluate Efficacy and Tolerability of the Association of Valsartan and Amlodipine Versus Amlodipine Alone in the Treatment of Essential Arterial Hypertension - Stages I and II (Mild to Moderate).
Brief Title: Comparative Study of Valsartan and Amlodipine Versus Amlodipine Alone in Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CVAL489ABR02
Record Dates: First submitted 2006-06-01; First posted 2006-06-05 (Estimated); Last update posted 2011-11-08 (Estimated); Status verified 2006-06

CONDITIONS: Hypertension
Keywords: valsartan; amlodipine; hypertension
MeSH Terms: conditions — Hypertension | interventions — Valsartan

INTERVENTIONS:
Drug: valsartan

SUMMARY:
The objective of this study is to evaluate efficacy, safety and tolerability of the valsartan+amlodipine association in patients with mild to moderate essential hypertension, in comparison to amlodipine alone.

Patients should have mild to moderate essential hypertension [grades 1 and 2 of WHO classification (8)]. The diastolic blood pressure threshold for inclusion in this study is 95 mmHg, as these patients are more likely to benefit from association therapy than patients with lower diastolic blood pressure.

For safety reasons, patients with severe hypertension (grade 3 of WHO classification) will not be included in this study. Moreover, patients developing severe hypertension (MSDBP > 110 mmHg and/or MSSBP > 180 mmHg) during the open-label treatment phase will be discontinued from the study.

ELIGIBILITY:
Incl- Patients with mild to moderate essential hypertension (grade 1 and 2 of WHO classification).

- Patients with essential diastolic hypertension measured by a standard aneroid or mercury column sphygmomanometer showing MSDBP > 95 mmHg and < 110 mmHg and MSSBP <180 mmHg.

Exclusion Criteria:

* Severe hypertension (grade 3 of WHO classification: DBP >= 110 mmHg and/or SBP ≥ 180 mmHg) or malignant hypertension.
* Inability to completely discontinue all antihypertensive medications safely for a period of at least 2 weeks as required by the protocol.
* Evidence of a secondary form of hypertension, such as coarctation of aorta, hyperaldosteronism, unilateral or bilateral renal artery stenosis, Cushing's disease, pheochromocytoma, polycystic kidney disease, etc.

Ages: 21 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2004-03; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the mean sitting diastolic blood pressure after 8 weeks

SECONDARY OUTCOMES:
Change from baseline in the mean sitting systolic blood pressure from baseline after 8 weeks
Adverse events after 8 weeks
Change from baseline in standing blood pressure and heart rate after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland